CLINICAL TRIAL: NCT00216515
Title: A Prospective, Open-labeled, Multicenter Study of Galantamine on the Attention and Frontal Function of the Patients With Dementia of Alzheimer Type
Brief Title: The Efficacy of Galantamine on the Attention and the Frontal Function of the Patients With Dementia of Alzheimer Type
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005047
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; galantamine; attention; executive function
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to assess the efficacy of galantamine on the attention of patients with Alzheimer's Disease, how an improvement of attention of Alzheimer's Disease patients affects their activities of daily living, and the global benefit of galantamine.

DETAILED DESCRIPTION:
Recent studies suggest that an attention deficit occurs at early stage of Alzheimer's disease and affects patients' activities of daily living. In other words, some patients without language or visuospatial dysfunction have severe impairment of activities of daily living, which might result from attention deficit. Another recent clinical study showed that galantamine is more effective in attention and vigilance of Alzheimer's disease patients than donepezil. The study hypothesis is that galantamine will improve attention and frontal executive function in Alzheimer's disease patients and is well-tolerated. 8 mg/day for the first 4 weeks, 16 mg for the next 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 50 years or older
* Alzheimer's disease according to the criteria of DSM-IV15, NINCDS-ADRDA16
* Measuring standard MMSE-K 10 to 26
* Patients who are literate
* Dementia patients being nursed by the family
* Patients who submitted written consent before entering into the clinical trial (the guardian consent is also effective)

Exclusion Criteria:

* If the patient was taking AChEI (Tacrine, Donepezil, Rivastigmine) to treat dementia, the patient can enter into this clinical trial as long as he/she has not taken the drug within 15 days of the beginning of the clinical trial
* Neurodegenerative diseases (e.g. Parkinson's disease, Pick's disease, Huntington's disease, Down syndrome)
* Dementia related to head trauma and dementia related to brain damage due to cerebral hypoxia (hypoxic brain damage after cardiopulmonary resuscitation, hypoxic brain damage after surgery, hypoxic brain damage due to addiction, hypoxic brain damage due to shock)
* brain tumor, nerve syphilis, meningitis, encephalitis, brain tumor
* amentia
* epilepsy
* major psychiatric patients such as major depression and schizophrenia
* treatment-resistant gastric and peptic ulcer
* patients with clinically serious hepatic, renal, lung, endocrinal or metabolic disease(thyroid, parathyroid, pituitary, renal failure, diabetes mellitus)
* patients complaining of severe difficulty in urination
* patients who have undergone heart surgery within 6 months or patients who experienced myocardial infarction, patients with untreated congestive heart failure, patients with severe disorders in the mitral valve or aortic valve
* patients who have once taken the investigational drugs within the past 1 month from the beginning day of the clinical trial
* patients with uncontrolled diabetes mellitus (if the patient is taking medication and consults the doctor on a regular basis, he/she can participate in this clinical trial)
* patients who experienced hypersensitivity or allergy by a cholinesterase inhibitor
* patients who have not given their consent to the clinical trial, patients who are judged inappropriate to participate in this clinical trial by the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Attention and Executive function: Visual CPT, Visual Span, Color Trail Making test, Stroop test

SECONDARY OUTCOMES:
Cognition: Mini-Mental Sate Examination-Korean version (MMSE-K);Activities of Daily living: Seoul- Instrumental Activities of daily livings (S-IADL);Behavior: NPI-Q;Global Change: Global Deterioration Scale (GDS)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.